CLINICAL TRIAL: NCT03325322
Title: Frailty, Inflammation, and Stem Cell Functionality in Chronic Kidney Disease
Brief Title: Inflammation and Stem Cells in Diabetic and Chronic Kidney Disease
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to lack of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, LaTonya J. Hickson, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 16-010521
Record Dates: First submitted 2017-10-12; First posted 2017-10-30 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Chronic Kidney Diseases; Diabetes Mellitus; Diabetic Nephropathies
Keywords: Frailty; Inflammation; Mesenchymal stem cell; Mesenchymal stromal cell
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Diabetic Nephropathies; Frailty; Inflammation | interventions — fisetin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Fisetin 20 mg/kg/day, orally for 2 consecutive days
  Interventions: Dietary Supplement: Fisetin
- Placebo (Placebo Comparator): Placebo capsules orally for 2 consecutive days
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Dietary Supplement: Fisetin — Flavonoid family
  Arms: Treatment
Drug: Placebo oral capsule — Placebo
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The proposed studies will examine the effect of fisetin on adipose tissue-derived mesenchymal stem/stromal cell function, kidney function, markers of inflammation, and physical function in individuals with advanced chronic kidney disease.

DETAILED DESCRIPTION:
The proposed studies will examine the effect of fisetin on adipose tissue-derived mesenchymal stem/stromal cell function, kidney function, markers of inflammation, and physical function in individuals with advanced chronic kidney disease, particularly diabetic kidney disease. This study will involve a single 2-day oral treatment regimen with fisetin or placebo. Study subjects will be randomized 2:1 to study drug or placebo. Study visits will consist of blood, urine, and abdominal wall skin and subcutaneous fat samplings in addition to testing of physical strength at given time points. Subjects will be followed for a total of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-80 years
* Chronic kidney disease estimated glomerular filtration rate (eGFR) 15-60 ml/min/1.73m2
* For the diabetic kidney disease (DKD) subgroup: Diabetes mellitus (on medication)

Exclusion Criteria:

* Hemoglobin A1c>11% at screening for the DKD subgroup
* Body weight >150 kg or body mass index>50
* Pregnancy
* Active glomerulonephritis treated with immunosuppressive therapy
* Solid organ transplantation (eg. kidney, pancreas, liver, lung, heart)
* Active immunosuppression therapy
* History of active substance abuse (including alcohol) within the past 2 years,
* Current alcohol abuse (>3 alcoholic beverages/day or >21 per week),
* Human immunodeficiency virus infection
* Active hepatitis B or C infection
* Total bilirubin >2x upper limit of normal
* Uncontrolled psychiatric disorder
* Uncontrolled systemic lupus erythematosus
* Uncontrolled pleural/pericardial effusions or ascites
* New invasive cancer except non-melanoma skin cancers
* Invasive fungal or viral infection
* Inability to tolerate oral medications
* Known hypersensitivity or allergy to Fisetin
* Subjects taking medications that are sensitive to substrates or substrates with a narrow therapeutic range for CYP3A4, CYP2C8, CYP2C9, or CYP2D6CYP2C9, CYP2C19, CYP1A2, Other (OATP1B1) (Unless willing and able to stop or modify the dosing of the drug) or strong inhibitors or inducers of CYP3A4 (e.g. cyclosporine, tacrolimus or sirolimus).
* Tyrosine kinase inhibitor therapy
* Subjects on therapeutic doses of anticoagulants (e.g., warfarin, heparin, low molecular weight heparin, factor Xa inhibitors, etc.).
* Subjects on full-dose 325 mg aspirin or other anti-platelet agents (eg. clopidogrel) daily who are unable or unwilling to reduce or hold therapy prior to and during the 2-day drug dosing. Subjects may continue their previous regimen on day 3.
* Baby aspirin (81 mg), if necessary for cardioprotection, will be allowed but encouraged to hold.
* Subjects taking proton pump inhibitors who are unable or unwilling to reduce or hold therapy 2 days prior to and during the 2-day drug dosing. Subjects taking H2-antagonists and unwilling to discontinue therapy for 2 weeks before and one week following enrollment. (See Appendix 4)
* Subjects taking glimepiride or glyburide for diabetes therapy who are unable or unwilling to reduce or hold therapy prior to and during the 2-day drug dosing.
* Subjects taking the following antimicrobial agents: Aminoglycosides, Azole antifungals (fluconazole, miconazole, voriconazole, itraconazole), Macrolides (clarithromycin, erythromycin), Antivirals (nelfinavir, indinavir, saquinavir, ritonavir, elbasvir/grazoprevir), Rifampin
* Corrected QT interval (QTc) >450 msec
* Tobacco use (smoking or chewing; Unless subject willing to reduce use by 50% prior to and during the study) - see Behavioral Modification information below.
* Inability to give informed consent
* Presence of any condition that the Investigator believes would put the subject at risk or would preclude the patient from successfully completing all aspects of the trial

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Change in inflammatory markers including C-reactive protein | 14 days
  To examine the effect of study drug (compared to placebo) on markers of inflammation in skin, fat, plasma, and urine measured at baseline and day 14
Effect on Mesenchymal stem cell function including cell migration | 14 days
  To examine the effect of study drug (compared to placebo) on mesenchymal stem cell function and vitality measured at baseline and day 14

SECONDARY OUTCOMES:
Effect on measures of Frailty including Fried Criteria | 4 months
  To examine the effect of study drug (compared to placebo) on markers of physical frailty (frailty phenotype).
Kidney function including estimated glomerular filtration rate | 4 months
  To examine the effect of study drug (compared to placebo) on kidney function.
Kidney function including urine protein excretion rate | 4 months
  To examine the effect of study drug (compared to placebo) on kidney function protein excretion
Number of participants with treatment-related adverse events including hospitalization | 12 months
  To assess the safety and tolerability of study drug taken over two days (compared to placebo)

CONTACTS AND LOCATIONS:
Overall Officials: LaTonya J Hickson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bian X, Snow ZK, Zinn CJ, Gowan CC, Conley SM, Bratulin AL, Elhusseiny KM, Miller J, Tchkonia T, Kirkland JL, Lerman LO, Hickson LJ. Activin A Antagonism with Follistatin Reduces Kidney Fibrosis, Injury, and Cellular Senescence-Associated Inflammation in Murine Diabetic Kidney Disease. Kidney360. 2025 Mar 28;6(8):1278-1291. doi: 10.34067/KID.0000000776. PMID 40152935
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials